CLINICAL TRIAL: NCT01952964
Title: The Effectiveness of a Physical Anti-microbial Spray Dressing in Preventing Tenckhoff Catheter Exit Site Infection for End Stage Renal Failure Patients
Brief Title: The Effects of Anti-microbial Spray Dressing in Preventing Tenckhoff Catheter Exit Site Infection for End Stage Renal Failure Patients
Acronym: JUCspray
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Queen Elizabeth Hospital (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TAM MEE LING BONNIE, Ms, The Queen Elizabeth Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KC/KE-10-0196/ER-3
Record Dates: First submitted 2013-09-25; First posted 2013-09-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Signs and Symptoms of Exit Site Infection; Physical Damage of the Tenckhoff Catheter; Skin Allery
Keywords: exit site infection; skin allergy; physical damage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- JUC spray dressing (Experimental)
  Interventions: Other: JUC spray dressing

INTERVENTIONS:
Other: JUC spray dressing — Intervention group Care of Tenckhoff catheter exit site using spray dressing. The detailed procedures will be introduced by the nurse according to the protocol of the unit. Please refer to Appendix III for details.
  Skin test with JUC spray will be carried out prior to the usage of JUC spray dressing for caring the exit site. For the first three days after patient has been discharged, study team members will perform telephone follow up. Patients are reminded to report for signs and symptoms of infection or physical damage of catheter noted. A routine follow up at the Renal Unit will be arranged at eight weeks intervals.

SUMMARY:
The present study aims to compare the differences in exit site infection between patients receiving spray dressing and conventional care. The outcome measures including catheter exit site infection rate, skin allergy, catheter damage and patient satisfaction

DETAILED DESCRIPTION:
Methods

The study will be conducted using randomized controlled trial.

Sampling

The subjects will be the patients with Tenckhoff Catheter recruited from the renal team in a regional acute hospital and a satellite dialysis centre. The sampling method will be convenience sampling. The subjects will be recruited sequentially after the insertion of Tenckhoff Catheter.

Inclusion criteria

* Patient with established Tenckhoff Catheter for at least 3 months
* Patient with skin condition healed satisfactorily

Exclusion criteria

* Patient presents with signs and symptoms of exit site infection e.g. purulent discharge, pain, and swab of exit cultured with positive growth.
* Patient with unhealed exit site.
* Patient currently requires antibiotics
* Patient shows sensitive to JUC Spray Dressing or 0.05% Chlorhexidine solution

(A) Control group Care of Tenckhoff catheter exit site using 0.05% Chlorhexidine solution (Guidelines on the care of peritoneal catheter exit site, Renal Unit, QEH). The detailed procedures will be introduced by the nurse according to the protocol of the unit. Please refer to Appendix II for details.

Skin test with 0.05% Chlorhexidine will be carried out prior to the usage of Chlorhexidine solution for caring the exit site. For the first three days after patient has been discharged, study team members will perform telephone follow up. Patients are reminded to report for signs and symptoms of infection or physical damage of catheter noted. A routine follow up at the Renal Unit will be arranged at eight weeks intervals.

(B) Intervention group Care of peritoneal catheter exit site using spray dressing. The detailed procedures will be introduced by the nurse according to the protocol of the unit. Please refer to Appendix III for details.

Data collection

Quantitative data collection such as demographic data, time of insertion of Peritoneal Catheter, history of allergy would be collected from patient's record. The condition of the exit site will be monitored daily by patient / carer. They are taught to report to the nurses for any abnormality noted such as signs and symptoms of infection, skin allergy and damage of the catheter. A comprehensive nursing assessment will be carried out at 8 weeks interval monthly for 6 months.

Data analysis

The data will be analyzed using PASW. The demographic data will be reported using means and standard deviation. Independent sample t-test will be used to compare the differences between groups. P<0.05 will be set as significant difference.

Ethical Considerations

All patients participate this study are on voluntary base. Before launching of the study, ethical approval from the Research Ethical Committee, The Hong Kong Polytechnic University and Ethical Committee, Kowloon Central Cluster will be obtained. A detailed explanation of the research objectives and different interventions will be provided to the patients verbally and in the information sheet. After passing the skin test on allergy reactions, patients agree to participate will need to sign the consent form.

During data collection, the research code will be assigned to each subject and the name will not be appeared on any research documentation to ensure confidentiality. The data will only be accessed by the research team members . Furthermore, the Research Ethical Committee (REC) and the Regulatory Authority of the study hospital will be granted direct access to the subject's study data for data verification. The Research Ethical Committee will spot check the clinical area during the study period to ensure research ethics are adhered and good clinical practices are maintained throughout the study.

ELIGIBILITY:
Inclusion Criteria:

- Patient with established Tenckhoff Catheter for at least 3 months with skin healed satisfactorily

Exclusion Criteria:

* Patient presents with signs and symptoms of exit site infection e.g. purulent discharge, pain, and swab of exit cultured with positive growth.
* Patient with unhealed exit site.
* Patient currently requires antibiotics
* Patient shows sensitive to JUC Spray Dressing or 0.05% Chlorhexidine solution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-09 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of spray dressing in preventing exit site infection | On going monitoring for six months
  sign and symptom of red, tenderness, hot and discharge.
Prevention of infection | Monitor the exit site for six months
  Exit site infection

SECONDARY OUTCOMES:
Prevention of skin allergy | 6 month monitoring
  Skin allergy

CONTACTS AND LOCATIONS:
Locations (1):
- Renal Unit of Queen Elizabeth Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Result] Davies SJ, Ogg CS, Cameron JS, Poston S, Noble WC. Staphylococcus aureus nasal carriage, exit-site infection and catheter loss in patients treated with continuous ambulatory peritoneal dialysis (CAPD). Perit Dial Int. 1989;9(1):61-4. PMID 2488184